CLINICAL TRIAL: NCT02930564
Title: The Challenge Study: A Dietary Personalization Protocol for Patients With Crohn's Disease and Deep Remission
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It is not possible to continue the study
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Arie Levine, Prof, Wolfson Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0186-16-WOMC
Record Dates: First submitted 2016-10-09; First posted 2016-10-12 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Glutens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a milk fat or gluten challenge (Experimental): patients will regress to the first stage diet with either a milk fat /emulsifier or a gluten/emulsifier challenge over 7 days.
  Interventions: Other: CDED + milk fat and gluten

INTERVENTIONS:
Other: CDED + milk fat and gluten — CDED phase 1- induction phase a milk fat /emulsifier challenge (one scoop of ice cream and one slice of yellow processed cheese every day in the evening over 7 days), or a gluten/emulsifier challenge ( 3-4 slices of bread)
  Other Names: Crohn's Disease Exclusion Diet (CDED)

SUMMARY:
The Challenge study is a prospective, open label, pilot trial in patients in deep remission on dietary maintenance therapy.

The purpose of this study is to determine whether they can consume some of the products that were eliminated from their diet, named the Crohn's Disease Exclusion Diet (CDED), and to evaluate if low dose exposure is harmful.

DETAILED DESCRIPTION:
The investigators have previously hypothesized that Crohn's disease may occur via a sequence of events involving dysbiosis and genetically determined or environmentally acquired defects in innate immunity, and have further hypothesized that the mechanism of EEN for induction of remission acts by reducing exposure to dietary components that may cause an acquired bacterial clearance defect or generate dysbiosis.

Based on this premise, the investigators developed a new exclusion diet. This diet, named the Crohn's Disease Exclusion Diet (CDED) reduces exposure to all the components identified in rodent models as well as two components that are highly suspect but have not been investigated in models. This diet was evaluated for induction of remission through week 12 and succeeded in inducing remission in 70% of 47 selected patients.

The investigators have now progressed to three randomized controlled trials to evaluate the diet in different populations with different disease severity, and the results from the first RCT demonstrate a high remission rate in the CDED arm. However , to date the investigators have used the same diet for all patients. The investigators are now encountering patients on the diet in deep remission, but the investigators do not know if they can consume some of the products ( such as milk fat and gluten) that were eliminated. The investigators therefore are starting to challenge our patients in deep remission with low dose exposure to evaluate if low dose exposure is harmful. The investigators wish to document this and obtain stool samples for calprotetctin and microbiome to investigate these patients at a microbiological level as well.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of Crohn's disease.
2. Patients in sustained remission with PCDAI 0 > 6 months
3. Ages 8-20
4. Normal CRP (CRP<0.5), normal Calprotectin (<100)
5. Patients with uncomplicated disease
6. Signed informed consent

Exclusion Criteria:

1. Patients with active disease (PCDAI >10)
2. Pregnancy
3. Patients with complicated disease (B2, B3)
4. Patients with recent onset use of an immunomodulator <12 weeks, or dose change in past 12 weeks.
5. Patients with current use of biologics.
6. Elevated CRP or Calprotetcin>100 at screening.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-05-29 (Actual); Study Completion 2022-05-29 (Actual)

PRIMARY OUTCOMES:
number of patients with calprotetctin elevation | day 14 or 21

CONTACTS AND LOCATIONS:
Overall Officials: Arie Levine, MD, Study Chair — Pediatric Gastroenterology and Nutrition Unit, The E. Wolfson MC, Tel-Aviv University, Holon, Israel
Locations (1):
- Wolfson Medical Center, Holon, Israel

IPD SHARING:
Plan to Share IPD: Undecided